CLINICAL TRIAL: NCT06179134
Title: Cognitive Rehabilitation Training for People With Multiple Sclerosis: a Randomized Controlled Trial
Brief Title: Cognitive Rehabilitation for People With Multiple Sclerosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Anthony Feinstein, Lead principal investigator, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-170
Record Dates: First submitted 2023-11-29; First posted 2023-12-21 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Multiple Sclerosis
Keywords: Cognitive rehabilitation; Goal Management Training
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled single-blinded trial with treatment and wait list control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cognitive rehabilitation group (Experimental): will be treated by GMT for 5 weeks (two hour sessions per week, one day of rest in between).
  Interventions: Behavioral: Goal Management Training
- wait-list control group (No Intervention): will be given a list cognitive compensatory strategies that they can do on their own to improve their memory.

INTERVENTIONS:
Behavioral: Goal Management Training — The main objective of GMT intervention are to train individuals to periodically "STOP "what they are doing, attend to task goals, evaluate their performance and monitor or check outcomes as they proceed (Levine & Stamenova, 2017).
  Arms: cognitive rehabilitation group

SUMMARY:
Cognitive rehabilitation is designed to enhance a person's capacity to process and interpret information and improve their ability to function in all aspects daily, family and community life. Given the clear and consistent documentation of cognitive deficits in persons with MS, the most notable deficit being information processing speed, learning and memory and executive function, there is an obvious need for effective cognitive rehabilitation.

The proposed study will be a randomized controlled single-blinded trial with treatment and wait-list control group. The treatment group will be administered the Goal Management Training (GMT) program; the wait-list control group will be given usual care by their neurologist.

Intervention details:

The treatment group will receive in-person computerized cognitive rehabilitation (using the GMT program) (virtual training is optional) for 5 weeks (40-min sessions, twice per week), session will be tailored according to patient cognitive concerns at index assessment, and level of ability.

The wait list control group, will not receive treatment

Our primary outcome is information processing speed, secondary aims include learning and memory, and executive function. The minimal assessment of cognitive function in MS (MACFIMS) will be utilized to assess cognitive function. Additionally, tertiary aims include the following patient reported outcomes (PROs) will be collected: the hospital anxiety and depression scale (HADS), the modified fatigue impact scale (MFIS), the multiple sclerosis impact scale (MSIS-29), and the European quality of life (EQ-5D-5L) scale, to capture level of depression and anxiety, fatigue, impact of MS and quality of life.

Cognitive performance of all patients in both groups will be assessed at baseline, immediate post-5-week assessment, and at post 6-month follow-up assessment. We hypothesized that, compared to persons in the wait-list group, the participants receiving the GMT intervention will demonstrate significant improvements across all cognitive measures.

The wait-list control group will be given the option to receive the GMT intervention after the 6 months follow-up is complete. The individuals in the treatment group, wishing to continue with the GMT program, will be given a referral by Dr. Feinstein to a GMT certified therapist.

DETAILED DESCRIPTION:
Background:

Multiple sclerosis (MS) is a chronic disabling disease of the central nervous system, with symptom onset commonly occurring between the ages of 20 to 40 years old; with females being at a higher risk of developing MS than men. Cognitive impairment (CI) in the last decade has been acknowledged as a prevalent core feature of the MS clinical picture, along with mobility issues. Cognitive impairment affects up to 44.5 % of people with relapsing remitting MS (RRMS), 79.4 % in secondary progressive MS (SP), and up to 91.3 % in people with primary progressive MS. The most prominent deficits reported being information processing speed, learning and memory and executive function. Cognitive decline has been found to directly affect the quality of life of people with MS, impacting participation in social activities, driving abilities, employment productivity, and task of daily living. Currently there is no approved medication for the treatment of CI in MS, patients and their clinicians are left with basically symptomatic treatments. In the last decade there has been an increase in developing non-pharmacological rehabilitation treatment to reverse or to at least slow down the progression of cognitive decline with cognitive rehabilitation.

KEYWORDS Learning and memory; executive function; information processing speed; Goal Management Training; multiple sclerosis.

Proposal and aims:

Cognitive rehabilitation (CR) is designed to enhance a person's capacity to process and interpret information and improve their ability to function in all aspects of family and community life. Given the clear and consistent documentation of cognitive deficits in persons with MS, there is an obvious need for effective cognitive rehabilitation. A leading cognitive rehabilitation program called Goal Management Training® (GMT), has been used as an effective treatment for a variety of patient populations, including traumatic brain injury, stroke, schizophrenia, attention deficit hyperactivity disorder and multiple sclerosis for the treatment of cognitive deficits specifically executive function, learning & memory, and information processing speed.

A doctoral dissertation completed by Nadine Richards (2013), under the supervision of Brian Levine, investigated the effectiveness of the GMT intervention for multiple sclerosis (MS) patients with impaired cognition; using a double-blinded randomized controlled trial, with treatment group employing the GMT intervention and the sham group employing a psycho-educational intervention. Twenty eight participants were recruited, and randomized; participants in the GMT intervention learned stepwise strategies ("Stop-State-Split") to keep track of their daily activities, which included mindfulness training to enhance attentional awareness and control. The results post-training, revealed that compared to the psycho-educational control group, the GMT group was associated with greater improvement on test of executive-attentional processes as well as functional task performance and observable cognitive functioning in daily life activities, with effects remaining visible at 6 months. As of date this remains the only study carried out on patients with MS using the GMT intervention.

To elaborate further the GMT program, is a standardized metacognitive rehabilitation program designed to improve cognition. The GMT program contains 20 hours of training, that include employing the following tools psychoeducation, narrative examples mindfulness practice, and assignments completed both between and within sessions. The main objectives of the GMT intervention is to train individuals to periodically "STOP" what they are doing, attend to task goals, evaluate their performance, and monitor or check their performance as they proceed. The current version of GMT as mentioned above consists of 20 hours of training and its material and manual were made commercially available in 2012 by Baycrest Hospital (https://gmt.learnworlds.com/). The GMT cognitive rehabilitation training program is not considered a medical device and therefore not subject to Health Canada certification for use. As of April 20, 2023, the Goal Management program is now widely available through TELUS health's AbilitiCBT platform, and for clients across Canada and the United States (TELUS Health, 2023).

Given the devastating effects of cognitive impairment on social functioning, occupational functioning and everyday life activities in people with MS (pwMS), the amelioration of cognitive deficits is likely to improve everyday functioning in pwMS, thus greatly reducing the impact of the disease on the lives of people with MS and the overall cost of the disease to society at large. Therefore, efforts to improve cognitive abilities in this population may result in significant improvements in overall quality of life (QOL). The currently proposed study seeks to do just that.

The proposed pilot study will be a randomized controlled single-blinded trial with treatment and wait list control group. We aim to assess information processing speed, learning and memory, and executive function. The minimal assessment of cognitive function in MS (MACFIMS) will be utilized, to assess cognitive function. Additionally, the following PROs will be collected: the hospital anxiety and depression scale (HADS), the modified fatigue impact scale (MFIS), the multiple sclerosis impact scale (MSIS-29), and the European quality of life - 5 dimension - 5 level (EQ-5D-5L) scale, in order to capture level of, depression and anxiety, fatigue, impact of MS and quality of life. Patients in the cognitive rehabilitation group will be treated by GMT for 5 weeks (2 hour sessions, twice per week). The wait list control group will be given usual care/ routine care which consist of being provided with a list of cognitive compensatory strategies to do on their own. Cognitive performance of all patients in both groups will be assessed at baseline, immediate post-5-week assessment, and at post 6 month follow-up assessment. We hypothesized that, compared to persons in the wait-list control group, the participants receiving the Goal Management Training would demonstrate significant improvements across all cognitive measures.

ELIGIBILITY:
Inclusion Criteria:

* A define diagnosis of multiple sclerosis (which will include clinically isolate syndrome, radiologically isolated syndrome and neuromyelitis optica spectrum disorder).
* A performance below 1.5 or 2 standard deviations (SD) compared to the normative mean in at least 20-30% of the test parameters.
* Corrected near vision of 20/70 or better (to see test material)

Exclusion Criteria:

* Exclude persons with a history of central nervous system disease other than MS
* Use of illicit drugs, phencyclidine (PCP), Lysergic acid diethylamide (LSD), stimulants, amphetamines, barbiturates, etc. (Cannabis use is accepted)
* Psychotic symptoms, bipolar disorder, schizophrenia
* Exclude persons who have used steroids within the past 3 months
* Exclude persons unable or unwilling to travel to the Centre or requires transportation by ambulance.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-03 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with improved Information processing speed | 5 weeks immediate post assessment, and 6 months post assessment
  The Symbol Digit Modality Test (SDMT), will be use to measure changes in processing speed. A poor SDMT score tells us that cognitive decline occurred.
  Scoring involves summing the number of correct substitutions within the 90 second interval (max = 110). Higher scores means a better outcome.

SECONDARY OUTCOMES:
Number of participants with improved learning and memory | 5 weeks immediate post assessment, and 6 months post assessment
  The California verbal learning test - 11 (CVLT-II) will be use to measure learning and memory.
  The CVLT-II is used to assess recall and recognition of items in a list of 16 nouns that belong to four categories (furniture, vehicles/ways of travelling, vegetables, and animals). the total raw score is the sum of correct responses on the five presentations. Higher scores means a better outcome.
Number of participants with improved executive function | 5 weeks immediate post assessment, and 6 months post assessment
  The Brief visuospatial memory test - revised (BVMT-R) will be use to measure executive function.
  Recall performance is recorded for each of the immediate recall trials (Trial 1, Trail 2, and Trial 3) and for the delayed recall trial (Delayed Recall).The recall scores are combined to form three additional summary measures of executive memory. Higher scores means a better outcome.

OTHER OUTCOMES:
Number of people with improved fatigue symptoms | 5 weeks immediate post assessment, and 6 months post assessment
  The Modified Fatigue Impact Scale (MFIS) will be administered to assess fatigue at each assessment.
  Items on the MFIS can be aggregated into three subscales (physical, cognitive, and psychosocial), as well as into a total MFIS score. All items are scaled so that higher scores indicate a greater impact of fatigue on a person's activities.
  The total MFIS score can range from 0 to 84. It is computed by adding scores on the physical, cognitive, and psychosocial subscales. A lower score means better outcome.
Number of participants with improved anxiety symptoms | 5 weeks immediate post assessment, and 6 months post assessment
  The Hospital Anxiety Depression Scale (HADS) will be administered.
  Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression. A lower score means a better outcome.
  0-7 = normal, 8-10 = borderline abnormal, and 11-21 = abnormal
Number of participants with improved depression symptoms | 5 weeks immediate post assessment, and 6 months post assessment
  The Hospital Anxiety Depression Scale (HADS) will be administered.
  Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression. A lower score means a better outcome.
  0-7 = normal, 8-10 = borderline abnormal, and 11-21 = abnormal

CONTACTS AND LOCATIONS:
Locations (1):
- Anthony Feinstein, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available on request from the corresponding author, Dr. Anthony Feinstein. The data are not publicly available due to restrictions e.g. their containing information that could compromise the privacy of research participants.

REFERENCES:
- [Background] Stamenova V, Levine B. Effectiveness of goal management training(R) in improving executive functions: A meta-analysis. Neuropsychol Rehabil. 2019 Dec;29(10):1569-1599. doi: 10.1080/09602011.2018.1438294. Epub 2018 Mar 14. PMID 29540124